CLINICAL TRIAL: NCT03064555
Title: Acute Physiological Response to Exercise in End Stage Renal Disease
Acronym: PRECISE
Status: Completed | Type: Observational
Sponsor: Coventry University (Other)
Responsible Party: Principal Investigator, Mr Scott McGuire, Clinical Exercise Physiologist (PhD), Coventry University
Other Study IDs: Acute Exercise Response, Renal
Record Dates: First submitted 2017-02-18; First posted 2017-02-27 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Renal Disease
Keywords: Renal; Acute; Exercise; Dialysis; Hemodialysis; End stage renal disease; Aerobic
MeSH Terms: conditions — Kidney Diseases; Motor Activity; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples Without DNA — Serum and plasma from whole blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with end stage renal disease: Cardiopulmonary exercise test
  Cardiopulmonary exercise testing will be conducted on an electronically braked cycle ergometer using a ramped protocol with participants being required to pedal until exhaustion.
  Constant load exercise test
  Constant load exercise will be performed for 30 min on an electronically braked cycle ergometer whilst seated in a dialysis chair. Blood sampling and echocardiogram will be measured throughout.
- Healthy participants: Cardiopulmonary exercise test
  Cardiopulmonary exercise testing will be conducted on an electronically braked cycle ergometer using a ramped protocol with participants being required to pedal until exhaustion.
  Constant load exercise test
  Constant load exercise will be performed for 30 min on an electronically braked cycle ergometer whilst seated in a dialysis chair. Blood sampling and echocardiogram will be measured throughout.

SUMMARY:
Chronic kidney disease (CKD) affects between 5-10% of the world's population, equating to ~740 million people worldwide. End stage renal disease (ESRD) is the result of a progressive loss of kidney function where the patient requires dialysis to replace the typical functions of the kidney. The quality of life of these individuals can be poor as a result of various complications associated with CKD (e.g. heart disease, diabetes, muscle wastage, decreased fitness). In an attempt to combat reduced physical fitness, many studies have applied long term exercise programmes. However, the body's response to exercise in people with CKD is not well understood and a set of guidelines that informs safe and effective exercise prescription is lacking.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) affects between 5-10% of the world's population, equating to ~740 million people worldwide. End stage renal disease (ESRD) is the result of a progressive loss of kidney function where the patient requires dialysis to replace the typical functions of the kidney. The quality of life (QOL) of these individuals is severely impaired as a result of various complications associated with CKD (e.g. heart disease, diabetes, muscle wastage, decreased fitness). In an attempt to combat this decrease in physical fitness, many studies have applied long term exercise interventions. However, the acute response to exercise in this population is not entirely understood and a comprehensive set of guidelines that informs safe and effective exercise prescription is lacking.

The use of exercise as a therapeutic intervention in ESRD has grown in popularity, and evidence provided by numerous long term studies indicates cardiopulmonary, metabolic and inflammatory system adaptations. Despite these positive findings, the specific mechanisms through which exercise benefits these patients have not yet been fully established. In addition, the extent to which 'normal' physiology is acutely altered by dialysis treatment, and the effect that aerobic exercise may have on this, is unknown.

In patients with ESRD, this study aims to characterise the acute physiological response to exercise under different conditions. In doing so, the study aims to inform the development of guidelines for safe and effective intra-dialytic exercise training.

ELIGIBILITY:
Participants with end stage renal disease

Inclusion criteria

* On hemodialysis for at least 3 months.
* 4 hours of dialysis 3 times per week.
* Urea reduction rate of at least 65% during the three months before enrolment.
* Age 18 years or older.
* Able to complete the CPEX and CLE test.

Exclusion criteria

* Clinically significant valvular insufficiency.
* Clinically significant dysrhythmia.
* Uncontrolled intra-dialytic blood pressure (systolic > 180, diastolic >95).
* Excessive fluid accumulation between dialysis sessions (>3 liters).
* Hemoglobin unstable (below 9.0 g/dL).
* Ischemic cardiac event (<1 month).
* Unable to exercise.
* Morbidly obese (BMI > 40).
* Clinically significant and still active inflammatory or malignant process.
* Planned kidney transplant during the duration of study.

Healthy participants

Inclusion criteria

* Age 18 years or older.
* Able to complete the CPEX and CLE test.

Exclusion criteria

* Significantly limiting disease or comorbidity which would prevent full participation in exercise testing or illicit an abnormal cardiorespiratory response to exercise.
* Chronic kidney disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with end stage renal disease:
  Patients will be recruited from the University Hospitals Coventry & Warwickshire hemodialysis unit identified by the research team and renal medical professionals.
  Healthy participants:
  Healthy participants will be recruited from Coventry University database of previous research participants. This group will comprise of 20 participants, age and weight matched to the patients with ESRD.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-09-23 (Actual)

PRIMARY OUTCOMES:
Gas analysis | 2 months
  Measurement of O2/CO2 kinetics.

SECONDARY OUTCOMES:
Echocardiogram | 2 months
  Measurement of regional wall motion abnormalities.
Echocardiogram | 2 months
  Measurement of ejection fraction.
Echocardiogram | 2 months
  Measurement of cardiac output.
Blood samples | 2 months
  Investigation of cardiac, inflammatory and hormonal response to exercise.
Non invasive cardiac output measurement (NICOM) | 2 months
  Measurement of cardiac output during exercise,

CONTACTS AND LOCATIONS:
Overall Officials: Dr Elizabeth Elizabeth, Study Director — Coventry University; Prof Derek Renshaw, Principal Investigator — Coventry University; Prof Alfonso Jimenez, Principal Investigator — Coventry University; Prof Nithya Krishnan, Principal Investigator — Coventry University
Locations (1):
- UHCW, Coventry, Warwickshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balady GJ, Arena R, Sietsema K, Myers J, Coke L, Fletcher GF, Forman D, Franklin B, Guazzi M, Gulati M, Keteyian SJ, Lavie CJ, Macko R, Mancini D, Milani RV; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Interdisciplinary Council on Quality of Care and Outcomes Research. Clinician's Guide to cardiopulmonary exercise testing in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 13;122(2):191-225. doi: 10.1161/CIR.0b013e3181e52e69. Epub 2010 Jun 28. No abstract available. PMID 20585013
- [Background] Gould DW, Graham-Brown MP, Watson EL, Viana JL, Smith AC. Physiological benefits of exercise in pre-dialysis chronic kidney disease. Nephrology (Carlton). 2014 Sep;19(9):519-27. doi: 10.1111/nep.12285. PMID 24899042
- [Background] Kettner A, Goldberg A, Hagberg J, Delmez J, Harter H. Cardiovascular and metabolic responses to submaximal exercise in hemodialysis patients. Kidney Int. 1984 Jul;26(1):66-71. doi: 10.1038/ki.1984.135. PMID 6482181
- [Background] Nelson A, Otto J, Whittle J, Stephens RC, Martin DS, Prowle JR, Ackland GL. Subclinical cardiopulmonary dysfunction in stage 3 chronic kidney disease. Open Heart. 2016 Feb 24;3(1):e000370. doi: 10.1136/openhrt-2015-000370. eCollection 2016. PMID 27127638
- [Background] Viana JL, Kosmadakis GC, Watson EL, Bevington A, Feehally J, Bishop NC, Smith AC. Evidence for anti-inflammatory effects of exercise in CKD. J Am Soc Nephrol. 2014 Sep;25(9):2121-30. doi: 10.1681/ASN.2013070702. Epub 2014 Apr 3. PMID 24700875
- [Background] Peres A, Perotto DL, Dorneles GP, Fuhro MI, Monteiro MB. Effects of intradialytic exercise on systemic cytokine in patients with chronic kidney disease. Ren Fail. 2015 Aug 14:1-5. Online ahead of print. PMID 26275117
- [Background] Cibulka R, Racek J. Metabolic disorders in patients with chronic kidney failure. Physiol Res. 2007;56(6):697-705. doi: 10.33549/physiolres.931128. Epub 2007 Feb 8. PMID 17298212
- [Result] Chapter 1: Introduction and definition of CKD-MBD and the development of the guideline statements. Kidney Int. 2009 Aug;76113:S3-8. doi: 10.1038/ki.2009.189. No abstract available. PMID 26746396